CLINICAL TRIAL: NCT02578992
Title: "Neutral Head Position" and "Head-lift Position" for Orotrachwal Intubation With "Trachway" Intubating Stylet in Adults
Brief Title: "Neutral Head Position" and "Head-lift Position" for Orotracheal Intubation With "Trachway" Intubating Stylet in Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tri-Service General Hospital (Other)
Responsible Party: Principal Investigator, Wei-Hung Chan, Dr., Tri-Service General Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2-103-05-125
Record Dates: First submitted 2015-10-13; First posted 2015-10-19 (Estimated); Results first posted 2016-12-09 (Estimated); Last update posted 2016-12-09 (Estimated); Status verified 2016-10

CONDITIONS: Intubation; Difficult
Keywords: intubating stylet; head and neck position

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Head-lift Position (Experimental): The patients' head was placed in the head-lift position(A 7 cm high pillow was set beneath the patients' head with head in neutral position) and then the patient was intubated with Trachway by single-handed chin lift technique
  Interventions: Procedure: Head-lift position; Device: 7cm high pillow
- Neutral Position (No Intervention): The patients' head was placed in the neutral position and then the patient was intubated with Trachway by single-handed chin lift technique

INTERVENTIONS:
Procedure: Head-lift position — A 7 cm high pillow was set beneath the patients' head with head in neutral position for intubation.
  Arms: Head-lift Position
Device: 7cm high pillow — A 7 cm high pillow was set beneath the patients' head with head in neutral position for intubation.
  Arms: Head-lift Position

SUMMARY:
The purpose of this study is to investigate two different patient's head and neck positions(neutral head position and head-lift position) for the effectiveness of orotracheal intubation with using the "Clarus Video System (Trachway®)" intubating stylet.

DETAILED DESCRIPTION:
The sniffing position has traditionally been considered the optimal head position for direct laryngoscopy, However, it may aggravate cervical spine injury. The Trachway® video stylet is an intubating device that may avoid cervical movement during intubation. Nonetheless, the effectiveness of limited neck movement in patients with neutral head or head-lift position using the Trachway® video stylet remains unclear. The purpose of this study was to compare the intubation time of the two positions with the Trachway® video stylet.

ELIGIBILITY:
Inclusion Criteria:

* patients scheduled for various surgeries requiring general anesthesia with tracheal intubation
* American Society of Anesthesiologists(ASA) physical status classification I-III

Exclusion Criteria:

* pneumothorax
* room air saturation by pulse oximeter saturation less than 96%
* vocal cord palsy
* craniofacial anomaly
* congenital upper airway anomaly
* upper airway disease
* cervical spine pathology
* head and neck tumor status post radiotherapy
* an increased risk of regurgitation or pulmonary aspiration
* a history of difficult tracheal intubation

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Actual)
Dates: Start 2014-12; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Tri-Service General Hospital, Taipei, Taiwan, Taiwan

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients aged 20-80 years who were scheduled for various surgeries requiring general anesthesia with tracheal intubation were recruited. All patients exhibited an American Society of Anesthesiologists physical status of I-III. From November 2014 to October 2015
Pre-assignment Details: Patient denied to participated, equipment unavailable or malfunction, difficult mask ventilation were excluded .
Groups:
- Head-lift Position: The patients' head was placed in the head-lift position(A 7 cm high pillow was set beneath the patients' head with head in neutral position). An assistant anesthesiologist standing beside the patient and opposite to the left of the head anesthesiologist performed the manual in-line stabilization to simulate the scenario of intubation in patients with cervical spine injury. Then the patient was intubated with Trachway by single-handed chin lift technique
  Head-lift position: A 7 cm high pillow was set beneath the patients' head with head in neutral position for intubation.
  7cm high pillow: A 7 cm high pillow was set beneath the patients' head with head in neutral position for intubation.
- Neutral Position: The patients' head was placed in the neutral position.An assistant anesthesiologist standing beside the patient and opposite to the left of the head anesthesiologist performed the manual in-line stabilization to simulate the scenario of intubation in patients with cervical spine injury. Then the patient was intubated with Trachway by single-handed chin lift technique
Period: Overall Study
Arm/Group | Head-lift Position | Neutral Position
Started | 65 (November 2014) | 65 (November 2014)
Completed | 62 (October 2015) | 62 (October 2015)
Not Completed | 3 | 3
Not completed — equipment not available or malfunction | 3 | 3

BASELINE CHARACTERISTICS:
Population: age from 20-80
Groups:
- Total: Total of all reporting groups
Arm/Group | Head-lift Position | Neutral Position | Total
Number analyzed (Participants) | 62 | 62 | 124
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.6 (14.8) | 50.0 (15.0) | 50.8 (14.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27 | 29 | 56
  Male | 35 | 33 | 68
Race/Ethnicity, Customized [Number; unit: participants]
  Asian | 62 | 62 | 124
Region of Enrollment [Number; unit: participants]
  Taiwan | 62 | 62 | 124
Height, Thyromental distance, Sternomental distance, Neck length [Mean (Standard Deviation); unit: cm]
  Height | 162.3 (8.8) | 161.9 (9.1) | 162 (9)
  Thyromental distance | 7.7 (1.1) | 8.0 (0.9) | 7.8 (1.0)
  Sternomental distance | 15.2 (1.9) | 15.7 (1.8) | 15.5 (1.8)
  Neck Length | 16.7 (1.8) | 17.3 (1.7) | 17.0 (1.7)
Body weight [Mean (Standard Deviation); unit: kilogram] | 66.08 (15.8) | 66 (12) | 66 (14)

OUTCOME MEASURES:

1. Primary Outcome: Intubation Time
Description: the interval from the intubating stylet touched the mouth to capnogram shown, with all attempts, and was recorded by an independent observer with a stop watch.
Time Frame: from the intubating stylet touched the mouth to the capnogram shown, up to 30 seconds, and the sum of all attempts
Measure: Median (Inter-Quartile Range); unit: seconds
Arm/Group | Head-lift Position | Neutral Position
Number analyzed (Participants) | 62 | 62
seconds | 17.5 [15 to 20] | 21 [19 to 23.25]

2. Secondary Outcome: Modified Cormack-Lehane Grade
Description: The laryngeal view was graded by the observer with modified Cormack-Lehane grade after epiglottis was identified on the video monitor.
  Scale range (1, 2, 3, 4). Grade 1 is considered to be a better outcome while grade 4 is considered to be a worse outcome.
Time Frame: during intubation, after epiglottis was identified on the video monitor
Measure: Mean (Full Range); unit: units on a scale
Groups:
- Neutral Head Position; Head-lift Position: The laryngeal view was graded by the observer with modified Cormack-Lehane grade after epiglottis was identified on the video monitor.
Arm/Group | Neutral Head Position | Head-lift Position
Number analyzed (Participants) | 62 | 62
units on a scale | 2.53 [1 to 4] | 1.83 [1 to 4]

3. Secondary Outcome: Mean Arterial Pressure
Description: compare the mean arterial pressure between two groups.
Time Frame: before and after intubation, up to 5 minutes
Measure: Mean (Standard Deviation); unit: mmHg
Groups:
- Neutral Head Position; Head-lift Position: Hemodynamic variables were recorded 3 min before, and 1, 3, and 5 min after intubation.
Arm/Group | Neutral Head Position | Head-lift Position
Number analyzed (Participants) | 62 | 62
mmHg | 82 (14) | 86 (12)

4. Secondary Outcome: Visual Analog Scale of Sore Throat
Description: All patients were asked to rate the degree of sore throat, using a visual analogue scale after anesthesia emergence in the post-anesthesia care unit.
  Scale range: 0-10. 0 is considered to be a better outcome while 10 is a worse outcome.
Time Frame: after anesthesia emergence 30 minutest, at post-anesthesia care unit
Measure: Mean (Full Range); unit: units on a scale
Groups:
- Neutral Head Position; Head-lift Position: All patients were asked to rate the degree of sore throat, using a visual analogue scale after anesthesia emergence in the post-anesthesia care unit
Arm/Group | Neutral Head Position | Head-lift Position
Number analyzed (Participants) | 62 | 62
units on a scale | 1.82 [0 to 10] | 1.73 [0 to 10]

ADVERSE EVENTS:
Time Frame: 1 day
Arm/Group | Head-lift Position | Neutral Position
Serious Adverse Events (participants affected / at risk) | 0/62 | 0/62
Other Adverse Events (participants affected / at risk) | 0/62 | 0/62

LIMITATIONS AND CAVEATS:
Tracheal intubation with Trachway was performed by an novice anesthesiologist.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No